CLINICAL TRIAL: NCT06219161
Title: The Acute Effect of a Theacrine-based Supplement on Mobilization of Various Stem Cell Populations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Compound Solutions Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: U0001
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Stem Cells

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double blind, crossover study with a two-week washout period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (NAD3) (Active Comparator): 344 mg microcrystalline cellulose,156 mg of a proprietary blend of Wasabia japonica (freeze-dried rhizome) cultivar, standardized to NLT 12,000 ppm isothiocyanates, 97.0% Theacrine, Copper Nicotinic Acid chelated complex (17-20% Copper by ICP-Mass spectroscopy) per capsule
  Interventions: Dietary Supplement: NAD3
- Placebo (Placebo Comparator): 500 mg of foodgrade mass, and color-matched microcrystalline cellulose per capsule
  Interventions: Dietary Supplement: NAD3

INTERVENTIONS:
Dietary Supplement: NAD3 — NAD3 supplement (per capsule): 344 mg microcrystalline cellulose,156 mg of a proprietary blend of Wasabia japonica (freeze-dried rhizome) cultivar, standardized to NLT 12,000 ppm isothiocyanates, 97.0% Theacrine, Copper Nicotinic Acid chelated complex (17-20% Copper by ICP-Mass spectroscopy)

SUMMARY:
The goal of the study is to determine the acute and short-term supplementation effect of a commercially available theacrine-containing supplement (NAD3) on numbers of various circulating stem cell populations in older adults.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled crossover study with 12 participants randomized to receive either NAD3® or a placebo for seven days. Blood samples are collected after an overnight fast, before and after the seven-day supplementation period, as well as one and two hours after the final supplement/placebo dose. Using flow cytometry, circulating stem cells, including lymphocytoid CD34+ stem cells (CD45dimCD34+), stem cells associated with vascular maintenance and repair (CD45dimCD34+CD309+), CD34+ stem cells linked to a progenitor phenotype (CD45dimCD34+CD309neg), circulating endothelial stem cells (CD45negCD31+CD309+), and mesenchymal stem cells (CD45negCD90+) are quantified.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 40-70
* BMI between 21-34.99 kg/m2
* Vital signs with in normal range (heart rate 60-100 beats/minute, blood pressure (40-44 years - 125/83, 45-49 years- 127/84, 50-54 years -129/85, 55-59 years - 131/86, >60 - 134/87), 36.4-37.4 degrees Celsius
* Sedentary to lightly active (2 or fewer days per week of exercise)

Exclusion Criteria:

* Female participants who are lactating, pregnant or planning to become pregnant during the study
* History of use of illicit drugs or other substances of abuse within 12 months of the screening visit (to be determined at screening)
* Tobacco during the 90 days prior to screening
* Current use of medication/dietary supplements that claim to or have an effect on age-related processes, e.g. "anti-aging" supplements. Participants must undergo a ≥7-day washout period of no supplementation to be eligible.
* Known allergy, intolerance or hypersensitivity to NAD3
* Self-reported active infection or illness of any kind
* Cognitively impaired and/or unable to give informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change of stem cell numbers in blood circulation. | Changes at 1 and 2 hours after consumption of study product.
  Flow cytometry evaluation of stem cell phenotype.

SECONDARY OUTCOMES:
Change to numbers of circulating HSC- CD45, CD34, CD133. | Changes at 1 and 2 hours after consumption of study product.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating CEC - CD45, CD31, CD309. | Changes at 1 and 2 hours after consumption of study product.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating MSC-CD45, CD31, CD90. | Changes at 1 and 2 hours after consumption of study product.
  Flow cytometry evaluation of stem cell phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States